CLINICAL TRIAL: NCT06393010
Title: The Effect of Online Rehabilitation Applications on Pain and Quality of Life in Textile Workshop Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Responsible Party: Principal Investigator, AYCAN ÇAKMAK REYHAN, Principal Investigator, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulBuuu
Record Dates: First submitted 2024-04-17; First posted 2024-05-01 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Musculoskeletal System Problems; Textile Worker; Tele-rehabilitation
Keywords: musculoskeletal system problems,; Textile worker; tele-rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise (Experimental): Participants in the research will undergo a three-week online rehabilitation program, three times a week, lasting 40-45 minutes each session. The program includes posture, stretching, joint range of motion, strengthening exercises, pain education, and discussions. Conducted via Zoom, only the practitioner will be present during sessions. Non-attendance for two consecutive sessions or failure to provide feedback will result in exclusion. Exercises cover various body areas and types, including posture correction, range of motion, stretching, isometric neck and shoulder exercises, stick exercises, and strengthening exercises.
  Interventions: Behavioral: online rehabilitation program
- plasebo (Experimental): They won't exercise. They will only be evaluated at the beginning and after 2 months.
  Interventions: Behavioral: online rehabilitation program

INTERVENTIONS:
Behavioral: online rehabilitation program — Participants in the research will undergo a three-week online rehabilitation program, three times a week, lasting 40-45 minutes each session. The program includes posture, stretching, joint range of motion, strengthening exercises, pain education, and discussions. Conducted via Zoom, only the practitioner will be present during sessions. Non-attendance for two consecutive sessions or failure to provide feedback will result in exclusion. Exercises cover various body areas and types, including posture correction, range of motion, stretching, isometric neck and shoulder exercises, stick exercises, and strengthening exercises.

SUMMARY:
Musculoskeletal problems are a common health issue among individuals working in textile workshops, attributed to factors such as ergonomic risks in working conditions, personal characteristics of employees, and other workplace factors. Neck pain, back pain, shoulder pain, wrist pain, hand and finger pain, knee pain, and foot pain are frequently observed issues among those working in textile workshops, negatively impacting their functionality and quality of life.

The research aims to investigate the effects of online rehabilitation education on pain and quality of life among textile workers. Participants aged between 21 and 52 working in textile workshops will be included in the study. All participants will be evaluated twice, before and after treatment, with all assessments conducted face-to-face. Demographic information such as age, gender, marital status, etc., will be assessed using a structured socio-demographic form. Pain levels will be assessed using the 100 mm VAS, quality of life will be assessed using the SF-36 questionnaire, and posture evaluation will be conducted using anterior and lateral posture analysis. The rehabilitation program administered to participants will take place over a period of 3 months, with sessions conducted three times a week on an online platform. The rehabilitation program will include posture exercises, stretching exercises, exercises for normal joint range of motion, strengthening exercises, regional pain education (shoulder, elbow, hip, wrist), and discussions on good and poor posture, lasting approximately 40-45 minutes.

DETAILED DESCRIPTION:
Musculoskeletal system problems are a common health issue among individuals working in textile workshops. The causes of these problems include ergonomic risks in working conditions, personal characteristics of employees, and other workplace factors. Ergonomic risks are the most significant cause of musculoskeletal system problems in textile workshops. These risks can stem from factors such as the working positions of employees, equipment used, and the nature of the work itself. For example, factors like prolonged static postures, lifting and carrying heavy objects, performing repetitive movements, and using poorly designed equipment can contribute to musculoskeletal system problems. Personal characteristics of employees can also increase the risk of musculoskeletal system problems. For instance, employees who start working at a young age, are overweight, have poor posture habits, or smoke are more susceptible to these problems. Other workplace factors can also contribute to musculoskeletal system problems. Factors like poor ventilation, noise, and lighting can adversely affect the musculoskeletal system of employees. These problems typically manifest with symptoms such as pain, loss of strength, numbness, tingling, and swelling. In some cases, they can lead to more serious issues such as muscle tears and osteoarthritis. Common problems among individuals working in textile workshops include neck pain, back pain, shoulder pain, wrist pain, hand and finger pain, knee pain, and foot pain. These problems negatively impact the functionality and quality of life of individuals working in textile workshops.

The aim of the research is to examine the impact of an online rehabilitation program applied to individuals working in textile workshops on pain and quality of life. The desired outcome of the research is for the online rehabilitation program applied to individuals working in textile workshops to reduce pain symptoms and increase their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 21 and 52. To have worked in the textile sector for at least 2 years. To be a smartphone user.

Exclusion Criteria:

* Having a surgical history in the past six months. Having a history of cardiovascular disease that would hinder exercise. Having mental disorders. Having received physical therapy in the past six months.

Ages: 21 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
VAS scale for pain assessment | baseline and 8 weeks assessment
  Participants' pain will be assessed using the 100 mm Visual Analog Scale (VAS) in the research conducted with individuals working in textile workshops. The participants' pain will be evaluated at three time intervals: at rest, while working in the textile workshop, and at night. Participants will be asked to mark their perceived pain intensity on a straight line of 0 mm (no pain at all) to 100 mm (unbearable pain). The intensity of the perceived pain will be measured and recorded in millimeters (mm) at the end of the assessment.

SECONDARY OUTCOMES:
Posture assessment | Baseline and 8 weeks assessment
  The posture of individuals employed in the textile workshop included in the study will be evaluated through anterior and lateral posture analysis.
SF36 scale for quality of life assessment | Baseline and 8 weeks assessment
  The quality of life of individuals employed in the textile workshop included in the study will be evaluated using the Short Form-36 (SF-36) scale. The scale includes questions related to physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, mental health, energy, pain, and general perception of health. Textile workers will choose the response option that best suits them from the questionnaire. The scale is scored between "0" and "100". A score of "0" indicates poor health status, while a score of "100" indicates no health problems.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Bilgi University, Istanbul, Turkey (Türkiye)